CLINICAL TRIAL: NCT00291746
Title: A Single-Blind Single Arm Study to Validate the Reflux Disease Questionnaire (RDQ) for the Diagnosis of Reflux Disease in Primary Care in Patients Treated With Esomeprazole 40 mg o.d.
Brief Title: Validation of RDQ Questionnaire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: D9914C00002; DIAMOND
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole
Procedure: Bravo technique

SUMMARY:
The primary objective of this study is to determine the accuracy of the Reflux Disease Questionnaire (RDQ) as a diagnostic test for gastroesophageal reflux disease. Symptom evaluation by the RDQ will be compared with other established approaches to the diagnosis of gastroesophageal reflux disease (GERD) in a primary care patient population with symptoms thought to be of upper gastrointestinal (GI) tract origin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who seek medical advice at their family doctor (primary care physician) for symptoms thought by the primary care physician to arise from the upper GI tract
* The symptoms thought to pertain to the upper GI tract must have been present for at least 4 weeks prior to Visit 1 and to have occurred at least twice a week during that period
* The symptoms thought to pertain to the upper GI tract must have been of at least mild severity for a minimum of 3 days during the week prior to Visit 1

Exclusion Criteria:

* Upper GI endoscopy performed within a year prior to Visit 1
* Previous anti-reflux surgery, surgery for peptic ulcer or any form of upper gastrointestinal resective surgery
* Contra-indication to the Bravo™ procedure such as subjects with a history of bleeding diathesis, strictures anywhere along the GI-tract, esophageal varices, obstructions, or subjects equipped with a pacemaker, an implantable cardiac defibrillator or an implantable neurostimulator (NB: subjects with severe esophagitis (grade D) confirmed by endoscopy at Visit 2 can continue the study without performing the Bravo™ procedure)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2005-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Selection of RDQ items (RDQ will be completed by subject at Screening and visit 4)
Presence/absence of GERD as assessed by endoscopic Los Angeles (LA) grade (gastroesophageal endoscopy will be performed at visit 2)
pH monitoring (% time with esophageal pH<4; Bravo pH-Monitoring will be performed from visit 2 to 3.1)
Symptom Associated Probability (outcome test for Bravo pH monitoring)
Outcome of PPI test (is assessed between visit 3.2 and 4.

SECONDARY OUTCOMES:
Mean item score for the GSRS dimensions at the initial and last visit (as assessed by answers of patient at visit 1 and visit 4)
RDQ item scores and RDQ mean item scores for RDQ dimensions at baseline and at the end of treatment (as assessed by answers of patient at Screening and visit 4)
Occurrence and severity of clinical symptoms at the initial and last visit (as reported by the subject)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (30):
- Canada (7):
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, North York, Ontario
  - Research Site, Mirabel, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Saint-Léonard, Quebec
- Denmark (4):
  - Research Site, Glostrup Municipality
  - Research Site, Herning
  - Research Site, Odense
  - Research Site, Randers
- Germany (10):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Garmisch-Partenkirchen
  - Research Site, Halle
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Münster
  - Research Site, Siegen
- Research Site, Bergen, Norway
- Sweden (4):
  - Research Site, Gothenburg, Västra Götaland County
  - Research Site, Lund
  - Research Site, Skövde
  - Research Site, Stockholm
- United Kingdom (4):
  - Research Site, Bicester
  - Research Site, Coventry
  - Research Site, London
  - Research Site, West Bromwich

REFERENCES:
- [Derived] Vakil N, Niklasson A, Denison H, Ryden A. Symptom profile in partial responders to a proton pump inhibitor compared with treatment-naive patients with gastroesophageal reflux disease: a post hoc analysis of two study populations. BMC Gastroenterol. 2014 Oct 10;14:177. doi: 10.1186/1471-230X-14-177. PMID 25304129
- [Derived] Bytzer P, Jones R, Vakil N, Junghard O, Lind T, Wernersson B, Dent J. Limited ability of the proton-pump inhibitor test to identify patients with gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1360-6. doi: 10.1016/j.cgh.2012.06.030. Epub 2012 Jul 17. PMID 22813439
- [Derived] Dent J, Vakil N, Jones R, Bytzer P, Schoning U, Halling K, Junghard O, Lind T. Accuracy of the diagnosis of GORD by questionnaire, physicians and a trial of proton pump inhibitor treatment: the Diamond Study. Gut. 2010 Jun;59(6):714-21. doi: 10.1136/gut.2009.200063. PMID 20551454